CLINICAL TRIAL: NCT02299024
Title: Prescribing Opioid Pain Relievers in the Emergency Department: Understanding and Optimizing the Encounter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Emergency Medicine Foundation (Other)
Responsible Party: Principal Investigator, Danielle McCarthy, Assistant Professor of Emergency Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SP0017808
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Opioid Use, Unspecified
Keywords: opioids; health literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Patients in this arm are discharged from the Northwestern Emergency Department with standard communication about their prescribed opioid pain medication from their care providers. They are called for a follow up survey 4-7 days after their visit.
- Dual Modality Educational Intervention (Experimental): Patients in this arm are discharged from the ED with an additional information sheet about their prescribed opioid pain medication, via the intervention titled "Additional Opioid Information". The sheet is read aloud to them by a research assistant. They are called 4-7 days later for a follow up survey.
  Interventions: Behavioral: Additional Opioid Information

INTERVENTIONS:
Behavioral: Additional Opioid Information — Patients receiving this intervention are given additional information about the opioid pain medication that they are receiving in the form of a one page handout. The hand out was written in a health-literacy appropriate manner. A research assistant read the handout to them out loud, and they were given a copy to take home with them.
  Arms: Dual Modality Educational Intervention

SUMMARY:
The investigators overall study objective is to improve patients knowledge and safe use of opioid pain relievers upon discharge from the Emergency Department.

DETAILED DESCRIPTION:
Recent studies indicate that emergency department (ED) discharge processes - including written and spoken communications - are inadequate, and patients often leave without the knowledge necessary to properly care for themselves. In the context of opioid pain relievers, this lack of knowledge is potentially dangerous, as patients may not possess the requisite knowledge for safe use of their medication or an awareness of the dangers of medication misuse.

The aim of this study was to evaluate the impact of an opioid information sheet and spoken counseling on patient knowledge about opioids and safe use behaviors. The investigators conducted a randomized controlled pilot test of a dual-modality educational intervention (written information sheet and spoken counseling about opioids) to assess if the intervention can increase patient knowledge about opioid pain relievers. These activities were intended to guide future modification of educational interventions and the future development of best practices for emergency physician spoken counseling about opioid pain relievers.

ELIGIBILITY:
Inclusion Criteria:

* prescribed an opioid pain reliever
* English Speaking

Exclusion Criteria:

* Non-English Speaking
* Clinically unstable, psychologically impaired or intoxicated as judged by the research staff member.
* Chronic opioid use, defined as daily or near daily use of opioid pain relievers for the past 90 days.
* admitted to hospital
* unable to complete follow up phone interview in 4 - 7 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Knowledge of medication name | 4-7 days
  The primary outcome was the patients ability to identify the medication name of their prescribed opioid pain reliever upon follow-up.

SECONDARY OUTCOMES:
Knowledge and counseling recall outcomes | 4-7 days
  In addition to the outcome of medication name patients were asked additional knowledge and recall questions including: active ingredients in the medication, knowledge about safe daily dose of acetaminophen, side effects, recall of counseling about activities to avoid (drinking alcohol, driving vehicle), knowledge about addictive potential of the medication.
Actual Use outcomes | 4-7 days
  Patients were queried about their home use of the medication including: pain score at home, average number of tabs per day, and satisfaction with pain reduction. Additionally they were asked about the timing of any alcohol consumption or driving in relation to the timing of medication dosing.
Response to the intervention | 4-7 days
  Patients in the intervention arm were asked how they liked the intervention using a series of question with a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle McCarthy, MD MS, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States